CLINICAL TRIAL: NCT05800431
Title: Efficiency of NESA Microcurrents on Quality of Life in Geriatric Patients
Brief Title: NESA Microcurrents on Quality of Life in Geriatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Clinical Professor, University of Las Palmas de Gran Canaria
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: QueeNesa
Record Dates: First submitted 2023-03-17; First posted 2023-04-05 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-04

CONDITIONS: Aging
Keywords: physical therapy modality; sleep disorders; Quality of Life
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The evaluators of all the results and the main caregivers of the participating patients will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Non-invasive Neuromodulation (Experimental): The non-invasive neuromodulation experimental group, made up of 20 participants, are treated 20 sessions with the NXSignal non-invasive neuromodulation device (NESA)
  Interventions: Device: Non-invasive neuromodulation through the Nesa device
- Control group (CG) (No Intervention): Conventional care will be performed without interrupting their normal activity.

INTERVENTIONS:
Device: Non-invasive neuromodulation through the Nesa device — patients receive non-invasive neurostimulation through the Nesa device
  Arms: Non-invasive Neuromodulation

SUMMARY:
In recent years, the population of older adults (MA) in the world has been increasing, due to the increase in life expectancy and the decrease in the fertility rate. The United Nations (UN) places Spain as the most aged country in the world in the year 2050, with 40% of its population over 60 years of age. There is evidence that quality of life in the elderly is associated with variables linked to physical and psychological health. Thus, for example, previous research indicates that perceived health and cognitive functioning influence the perception of quality of life.

The NESA XSIGNAL® device is a low-frequency, non-invasive neuromodulation device that uses microcurrents to restore electrical balance in the body. This technology is approved as medical equipment and is CE marked.

This non-invasive neuromodulation equipment is starting to have promising results in patients with sleep disorders. So it can be a useful tool to reduce the impact on the geriatric patient's quality of life.

DETAILED DESCRIPTION:
The main objective will be to evaluate the efficacy of the application of non-invasive neuromodulation in the treatment of geriatric patients for the improvement of health-related quality of life. For this purpose, the investigators propose to carry out an interventional study with a sample of approximately 40 participants. Data will be recorded for 1 month and a half for each participant.

It is estimated 7 months from the design, management and development of the project, and it does not have sources of financing.

ELIGIBILITY:
Inclusion Criteria:

* Patients residing in the social-health care center under study.
* Stable medical and pharmacological condition.
* No cognitive impairment or mild cognitive impairment.

Exclusion Criteria:

* Patients with some of the contraindications for treatment with NESA device: pacemakers, internal bleeding, not applying electrodes on skin in poor condition, with ulcerations or wounds, acute febrile processes, acute thrombophlebitis and/or phobia of electricity,
* Not having signed the informed consent form.
* Patients with severe cognitive impairment, patients with severe cognitive impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Change in sleep quality | Measurement of change: before treatment (baseline), at two months (end of treatment), and at 6 months of treatment (follow-up period)
  The investigators want to see if there are improvements in the quality, efficiency, and quantity of sleep. The Pittsburgh Sleep Quality Index (PSQI) will be combined to report changes in the patient's sleep quality.
  Each of the sleep components yields a score ranging from 0 to 3, with 3 indicating the greatest dysfunction. The sleep component scores are summed to yield a total score ranging from 0 to 21 with the higher total score (referred to as global score) indicating worse sleep quality.
  Adding up the average scores of the seven factors gives a global PSQI score from 0 to 21, with 0-4 indicating "good" sleep and 5-21 indicating "poor" sleep
Change in quality of life | Measurement of change: before treatment (baseline), at two months (end of treatment), and at 6 months of treatment (follow-up period)
  The investigators want to see if the quality of life of patients improves when their relatives receive treatment. The Spanish version of the World Health Organization Quality of Life of Older Adults (WHOQOL-OLD) scale will be used.
  The WHOQOL-OLD is made up of 24 Likert-type scale items divided into six areas Likert-type scale, divided into six areas: sensory skills, autonomy, past activities abilities, autonomy, past, present and future activities, social participation, death and intimacy. Each of these areas contains four items, with a final score ranging from 4 to 20, provided that all items in the same area have been completed. The higher the score, the better the quality of life in each area.
Changes in mood | Measurement of change: before treatment (baseline), at two months (end of treatment), and at 6 months of treatment (follow-up period)
  The investigators will use the Geriatric Depression Scale (GDS).
  This is a questionnaire for screening for depression in people over 65 years of age. The main caregiver must answer 15 questions, one point is assigned for each answer that matches the one reflected on the side (affirming depression). The cut-off points are:
  * normal: 0 to 5 points
  * moderate depression: 6 to 10 points;
  * severe depression: more than 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: Aníbal Báez Suárez, PhD, Principal Investigator — University of Las Palmas de Gran Canaria
Locations (1):
- Aníbal Báez Suárez, Las Palmas de Gran Canaria, Spain, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogawa T, Koike M. Independent factors that attenuate the effectiveness of fracture rehabilitation in improving activities of daily living in female patients aged 80 years and above. Aging Clin Exp Res. 2022 Apr;34(4):793-800. doi: 10.1007/s40520-021-01992-y. Epub 2021 Oct 8. PMID 34623628
- [Background] Gottschalk S, Konig HH, Schwenk M, Nerz C, Becker C, Klenk J, Jansen CP, Dams J. Cost-Effectiveness of a Group vs Individually Delivered Exercise Program in Community-Dwelling Persons Aged >/=70 Years. J Am Med Dir Assoc. 2022 May;23(5):736-742.e6. doi: 10.1016/j.jamda.2021.08.041. Epub 2021 Oct 7. PMID 34626579
- [Background] Tang T, Jiang J, Tang X. Psychological risk and protective factors associated with depression among older adults in mainland China: A systematic review and meta-analysis. Int J Geriatr Psychiatry. 2022 Jan;37(1). doi: 10.1002/gps.5637. Epub 2021 Oct 14. PMID 34633701
- [Background] Coin A, Devita M, Trevisan C, Biasin F, Terziotti C, Signore SD, Fumagalli S, Gareri P, Malara A, Mossello E, Volpato S, Monzani F, Bellelli G, Zia G, Ranhoff AH, Antonelli Incalzi R. Psychological Well-Being of Older Adults With Cognitive Deterioration During Quarantine: Preliminary Results From the GeroCovid Initiative. Front Med (Lausanne). 2021 Sep 22;8:715294. doi: 10.3389/fmed.2021.715294. eCollection 2021. PMID 34631737